CLINICAL TRIAL: NCT01085097
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability and Clinical Effect of Laquinimod in Active Lupus Nephritis Patients, in Combination With Standard of Care (Mycophenolate Mofetil and Steroids)
Brief Title: A Study of Laquinimod in Participants With Systemic Lupus Erythematosus (SLE) Active Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LN-LAQ-201; 2010-018329-20 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-11 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Lupus Nephritis
Keywords: Systemic Lupus Erythematosus (SLE); Lupus Nephritis; Laquinimod
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — laquinimod; Mycophenolic Acid; Prednisolone; Prednisone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 2 capsules of placebo matching to laquinimod orally once daily (QD) for 24 weeks, MMF 500 mg tablet orally twice daily (BID) for the first week then 1 gram (g) BID from Week 2 to Week 28, and MP 500 mg/day intravenously (IV) from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which is tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Prednisolone/Prednisone; Drug: Placebo; Drug: Methylprednisolone
- Laquinimod 0.5 mg (Experimental): Participants will receive 1 capsule of laquinimod 0.5 mg and 1 capsule of placebo matching to laquinimod orally QD for 24 weeks, MMF 500 mg tablet orally BID for the first week then 1 g BID from Week 2 to Week 28, and MP 500 mg/day IV from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which is tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
  Interventions: Drug: Laquinimod; Drug: Mycophenolate Mofetil; Drug: Prednisolone/Prednisone; Drug: Placebo; Drug: Methylprednisolone
- Laquinimod 1 mg (Experimental): Participants will receive 2 capsules of laquinimod 0.5 mg orally QD for 24 weeks, MMF 500 mg tablet orally BID for the first week then 1 g BID from Week 2 to Week 28, and MP 500 mg/day IV from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which is tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
  Interventions: Drug: Laquinimod; Drug: Mycophenolate Mofetil; Drug: Prednisolone/Prednisone; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Laquinimod — Laquinimod will be administered per dose and schedule specified in the arm description.
  Arms: Laquinimod 0.5 mg; Laquinimod 1 mg
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil (MMF) will be administered per dose and schedule specified in the arm description.
Drug: Prednisolone/Prednisone — Prednisolone/Prednisone will be administered per dose and schedule specified in the arm description.
Drug: Placebo — Placebo matching to laquinimod will be administered per schedule specified in the arm description.
  Arms: Laquinimod 0.5 mg; Placebo
Drug: Methylprednisolone — Methylprednisolone (MP) will be administered per dose and schedule specified in the arm description.

SUMMARY:
The study aims to evaluate the safety and clinical effect of daily oral treatment with laquinimod capsules in active lupus nephritis participants. This study will assess Laquinimod doses of 0.5 milligrams (mg)/day and 1 mg/day in combination with standard of care treatment (mycophenolate mofetil [MMF] and corticosteroids). Laquinimod is a novel immunomodulating drug which is currently in advanced stages of development by Teva Pharmaceuticals Ltd. for Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with SLE
* Kidney biopsy within 12 months prior to baseline with a histological diagnosis of proliferative or membranous Lupus Nephritis (LN)
* Clinically active Lupus Nephritis as evident by urine protein-to-creatinine ratio (UPCR) of 1 or higher, for LN classes III, IV, or class V in combination with classes III or IV, or a UPCR of 2 or higher for LN class V, at screening or any time between screening and baseline.

Exclusion Criteria:

* Participants with severe renal impairment or dialysis
* Participants with a clinically significant or unstable medical or surgical condition
* Women who are pregnant or nursing or who intend to be during the study period
* Women of child-bearing potential who do not practice an acceptable method of birth control NOTE: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2012-10-24 (Actual); Study Completion 2012-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (30):
- United States (14):
  - Teva Investigational Site 1032, Phoenix, Arizona
  - Teva Investigational Site 1024, La Jolla, California
  - Teva Investigational Site 1028, Los Angeles, California
  - Teva Investigational Site 1025, San Leandro, California
  - Teva Investigational Site 1031, Baltimore, Maryland
  - Teva Investigational Site 1021, Rochester, Minnesota
  - Teva Investigational Site 1022, Lake Success, New York
  - Teva Investigational Site 1018, Manhasset, New York
  - Teva Investigational Site 1019, New York, New York
  - Teva Investigational Site 1017, New York, New York
  - Teva Investigational Site 1020, Charlotte, North Carolina
  - Teva Investigational Site 1016, Columbus, Ohio
  - Teva Investigational Site 1030, Charleston, South Carolina
  - Teva Investigational Site 1026, Chattanooga, Tennessee
- Canada (3):
  - Teva Investigational Site 1115, Edmonton, Alberta
  - Teva Investigational Site 1114, Winnipeg, Manitoba
  - Teva Investigational Site 1113, Toronto, Ontario
- France (2):
  - Teva Investigational Site 3510, Lille
  - Teva Investigational Site 3509, Paris
- Russia (6):
  - Teva Investigational Site 5006, Kazan'
  - Teva Investigational Site 5007, Kemerovo
  - Teva Investigational Site 5001, Moscow
  - Teva Investigational Site 5003, Moscow
  - Teva Investigational Site 5002, Moscow
  - Teva Investigational Site 5005, Yaroslavl
- United Kingdom (5):
  - Teva Investigational Site 3413, Birmingham
  - Teva Investigational Site 3409, Cambridge
  - Teva Investigational Site 3412, Dudley
  - Teva Investigational Site 3410, London
  - Teva Investigational Site 3411, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 2 capsules of placebo matched to laquinimod orally once daily (QD) for 24 weeks, mycophenolate mofetil (MMF) 500 milligrams (mg) tablet orally twice daily (BID) for the first week then 1 gram (g) BID from Week 2 to Week 28, and methylprednisolone (MP) 500 mg/day intravenously(IV) from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which was tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
- Laquinimod 0.5 mg: Participants received 1 capsule of laquinimod 0.5 mg and 1 capsule of placebo matched to laquinimod orally QD for 24 weeks, MMF 500 mg tablet orally BID for the first week then 1 g BID from Week 2 to Week 28, and MP 500 mg/day IV from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which was tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
- Laquinimod 1 mg: Participants received 2 capsules of laquinimod 0.5 mg orally QD for 24 weeks, MMF 500 mg tablet orally BID for the first week then 1 g BID from Week 2 to Week 28, and MP 500 mg/day IV from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which was tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
Period: Overall Study
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Started | 15 | 16 | 15
Received at Least 1 Dose of Study Drug | 15 | 16 | 15
Completed | 13 | 16 | 13
Not Completed | 2 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Treatment failure | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants randomly assigned to treatment. In this population, treatment was assigned based on the treatment to which participants were randomly assigned, regardless of which treatment they actually received.
Groups:
- Placebo: Participants received 2 capsules of placebo matched to laquinimod orally QD for 24 weeks, MMF 500 mg tablet orally BID for the first week then 1 g BID from Week 2 to Week 28, and MP 500 mg/day IV from Days 1 through 3, followed by oral prednisolone/prednisone (initial dose 40 mg/day which was tapered to 10 mg/day or less by the end of Week 20, on a fixed steroid-tapering regimen) from Day 4 through Week 28.
- Total: Total of all reporting groups
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (10.9) | 35.3 (11.5) | 32.7 (9.7) | 33.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 13 | 34
  Male | 4 | 6 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 1 | 3
  Black or African American | 3 | 4 | 1 | 8
  White | 7 | 11 | 9 | 27
  Hispanic | 2 | 1 | 4 | 7
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 28
Population: Safety analysis set included all randomly assigned participants who received at least 1 dose of study drug. In this set, participants were assigned to the treatment actually received, regardless of the assigned treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Number analyzed (Participants) | 15 | 16 | 15
participants | 14 | 15 | 15

2. Primary Outcome: Percent Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 24
Description: Estimated Glomerular Filtration Rate (eGFR) was calculated using the Modification of Diet in Renal Disease (MDRD) formula.
Time Frame: Baseline, Week 24
Population: Modified intent-to-treat (mITT) analysis set included all randomized participants, excluding observations after treatment failure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
Number analyzed (Participants) | 15 | 16 | 15
percent change | 12.1 (20.17) | 18.0 (30.65) | 24.3 (28.84)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: Safety analysis set included all randomly assigned participants who received at least 1 dose of study drug. In this set, participants were assigned to the treatment actually received, regardless of the assigned treatment.
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 1/15
Serious Adverse Events (participants affected / at risk) | 4/15 | 4/16 | 4/15
Other Adverse Events (participants affected / at risk) | 14/15 | 13/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Laquinimod 0.5 mg (N=16) | Laquinimod 1 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Laquinimod 0.5 mg (N=16) | Laquinimod 1 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushing's Syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gingival Recession (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema Peripheral (General disorders) | 4 (6) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (5)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 2 (3) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 4 (5) | 2 (2)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bacterial Test Positive (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood Albumin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Urea Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Weight Increased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Macroamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Burning Sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (6) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Affect Lability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (3) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vasectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.